CLINICAL TRIAL: NCT00538915
Title: Open Label, Phase III Safety, Efficacy, and Pharmacokinetic Study of NABI-IGIV 10% [Immune Globulin Intravenous (Human), 10%] in Subjects With Primary Immune Deficiency Disorders (PIDD)
Brief Title: Open Label, Phase III Study of NABI-IGIV 10% [Immune Globulin Intravenous(Human), 10%] In Subjects With Primary Immune Deficiency Disorders (PIDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nabi-7101
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2012-02

CONDITIONS: Primary Immune Deficiency Disorders (PIDD)
Keywords: immunodeficiency; humoral immunity; antibody deficiency; PID; PIDD
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immunologic Deficiency Syndromes | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nabi-IGIV Infused Every 3- or 4-Weeks (Experimental)
  Interventions: Biological: Nabi-IGIV 10% [Immune Globulin Intravenous (Human). 10%]

INTERVENTIONS:
Biological: Nabi-IGIV 10% [Immune Globulin Intravenous (Human). 10%] — Nabi-IGIV 10% [Immune Globulin Intravenous (Human), 10%] is a clear or slightly opalescent, colorless to pale yellow sterile solution of 10% protein concentration of immunoglobulin G (100mg/mL). It is packaged as 5g in 50mL solution and 10g in 100mL solution. Dosing will be 300-800 mg/kg based on subject's prior dosing history. Infusions will be every 3 or 4 weeks.

SUMMARY:
The purpose of this study is to determine if NABI-IGIV (10%) [Immune Globulin Intravenous (Human), 10%] is safe and effective in preventing serious bacterial infections (SBIs) in the treatment of patients with primary immune deficiency disorders (PIDD) when compared to historical control data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 6 and ≤ 75, with a documented and confirmed pre-existing diagnosis of chronic primary immune deficiency (PIDD) with a low total immunoglobulin G (IgG) level and deficient antibody production before chronic therapy (i.e., X-linked agammaglobulinemia, common variable immunodeficiency (CVID), Hyper IgM Syndrome with immunoglobulin G (IgG) deficiency, etc).
* Currently on immune globulin intravenous (IGIV) replacement therapy at a fixed interval and dosage with a total monthly dose of immune globulin intravenous (IGIV) between 300 and 800 mg/kg that has been stable for at least 3 months prior to screening.
* Documented (within 3 months) plasma immunoglobulin G (IgG) trough level of >500 mg/dL on current immunoglobulin G (IgG) therapy [immunoglobulin G (IgG) levels may be obtained at screening if previous results not available].
* Medical records documenting infections and treatment within the previous 2 years need to be available for review.
* Subject or legal guardian(s) must have given written informed consent/assent.
* If a menstruating female, have a negative serum or urine pregnancy test within 7 days prior to the first dose of Nabi-IGIV [immune globulin intravenous (Human) 10%] and agree to use an acceptable method of contraception or be at least one year post-menopausal or surgically sterile.

Exclusion Criteria:

* Received any blood product [other than immune globulin intravenous (IGIV)] within the last 3 months prior to screening or received any investigational agent [other than immune globulin intravenous (IGIV)] within the last four weeks prior to receiving Nabi-IGIV [immune globulin intravenous (Human) 10%].
* Known history of medically significant adverse reactions to other immunoglobulin G (IgG) or blood products.
* Known selective immunoglobulin A (IgA) deficiency, history of allergic reaction to products containing immunoglobulin A (IgA) or has a history of antibodies to immunoglobulin A (IgA).
* Known significant proteinuria and/or has a history of acute renal failure/or severe renal impairment [blood urea nitrogen (BUN) or creatinine more than 1.5 times the upper limit of normal].
* Known history or current diagnosis of deep venous thrombosis.
* Known medical condition that is known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, human immunodeficiency virus (HIV) infection, acquired immunodeficiency syndrome (AIDS), or chronic or recurrent neutropenia (absolute neutrophil count less than 500 mm3).
* Current daily use of corticosteroids (> 10 mg of prednisone equivalent /day for > 30 days), immunosuppressants or immunomodulators. (Intermittent corticosteroid use during the study is allowable, if medically necessary.)
* Known non-controllable arterial hypertension (systolic blood pressure (BP) > 160 mmHg and /or diastolic BP >100 mmHg.)
* Known anemia at screening (hemoglobin <10 g/dL).
* Subject is pregnant or lactating.
* Known history of illicit drug use within 3 months prior to the administration of the investigational product and for the study duration.
* Have any condition judged by the study physician to preclude participation in the study, including any psychological disorder, which might hinder compliance.
* Known active viral or bacterial infection or symptoms/signs consistent with such an infection within the two weeks prior to the initial dose of investigational product infusion. Subjects may be on antibiotics as long as signs/symptoms of infection have been absent for two weeks prior to the initial infusion of investigational product (IP).
* Expectation of non-compliance with the protocol procedures and visit schedule.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shailesh Chavan, M.D., Study Director — Biotest Pharmaceuticals Corporation
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Precision Trials LLC, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - 1st Allergy and Clinical Resaerch center, Centennial, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Marietta Pulmonary Medicine, Marietta, Georgia
  - Rush University Medical center, Chicago, Illinois
  - South Bend Clinic LLP, South Bend, Indiana
  - Kentuky Lung Clinic, PSC, Hazard, Kentucky
  - Institute For Allergy & Asthma, Wheaton, Maryland
  - Cardinal Glennon Children's MC, St Louis, Missouri
  - Women's and Children's Hospital of Buffalo, Buffalo, New York
  - University Hospital Case medical center, Cleveland, Ohio
  - Allergy/Immunology Research Center of north Texas, Dallas, Texas
  - AARA Research, Dallas, Texas
  - Allergy, Asthma & Immunology Clinic, PA, Irving, Texas
  - Bellingham Asthma, Allergy Clinic, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 24 September 2007. Last subject completed: 24 July 2009. 15 investigative sites, hospital clinics and private physician clinics.
Pre-assignment Details: This was an open study. All enrolled subjects received study medication.
Groups:
- Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval: Each subject received a total Nabi-IGIV 10% [Immune Globulin Intravenous (Human), 10%] infusion of 300-800 mg/kg per month administered intravenously every 3 or 4 weeks for approximately 1 year.
Period: Overall Study
Arm/Group | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval
Started | 63
Completed | 52
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 42
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Rate of Serious Bacterial Infections (SBIs) Per Person-year on Treatment
Description: Serious bacterial infections (SBIs) rate per person-years, including bacteremia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia and visceral abscess.
Time Frame: One year
Population: 63 subjects enrolled, received treatment and included in the Safety population. 5 subjects excluded from the Intent To Treat (ITT) population due to significant, excessive protocol violations and an insufficient number of infusions to elicit the intended effect.
Measure: Number; unit: SBIs Per Total Person-Years
Groups:
- Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval: Each subject received a total Nabi-IGIV 10% [Immune Globulin Intravenous (Human), 10%] infusion of 300-800 mg/kg administered intravenously every 3 or 4 weeks for approximately 1 year.
Arm/Group | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval
Number analyzed (Participants) | 58
SBIs Per Total Person-Years | 0.035

ADVERSE EVENTS:
Time Frame: An event was only included in the analysis of Adverse Events (AEs) if it had an onset date between the first administration of study drug and 28 days after the last administration of study drug, inclusive.
Arm/Group | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval
Serious Adverse Events (participants affected / at risk) | 7/63
Other Adverse Events (participants affected / at risk) | 47/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval (N=63)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Obstructive Chronic Bronchitis With Acute Exacerbation (Infections and infestations) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nabi-IGIV 10% Administered On A 3-Week or 4-Week Interval (N=63)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (10)
Fatigue (General disorders) | 15 (62)
Infusion Site Reaction (General disorders) | 5 (6)
Sinusitis (Infections and infestations) | 5 (5)
Blood Pressure Increased (Investigations) | 4 (5)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 27 (147)
Lethargy (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less